CLINICAL TRIAL: NCT00001371
Title: A Pilot Study of Topical Antiflammin-2 for Psoriasis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940048; 94-C-0048
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-12

CONDITIONS: Psoriasis
Keywords: Inflammation; Lipocortin; Phospholipase A-2; Skin; Uteroglobin; Psoriasis
MeSH Terms: conditions — Psoriasis; Inflammation

SUMMARY:
This study is a pilot trial designed to evaluate topical antiflammin-2, a phospholipase A2 (PLA2) inhibitor, in the treatment of chronic plaque psoriasis. Antiflammin-2 in an ointment base, or the vehicle alone will each be applied four times per day to a single plaque in a randomized, double-blinded fashion.

DETAILED DESCRIPTION:
This study is a pilot trial designed to evaluate topical antiflammin-2, a phospholipase A2 (PLA2) inhibitor, in the treatment of chronic plaque psoriasis. Antiflammin-2 in an ointment base, or the vehicle alone will each be applied four times per day to a single plaque in a randomized, double-blinded fashion.

ELIGIBILITY:
Patients must be age 18 or older.

Patients male or female must use contraception if of childbearing age. No men and women actively attempting to conceive a child during the time of drug testing. No pregnant or nursing women.

Patients must be otherwise healthy, immunocompetent, ambulatory patients with psoriasis who have more than 5 percent of their body surface area involved with the disease or who have localized disabling psoriasis.

Have failed one prior topical treatment regimen including topical cortiscosteroids, coat tar preparations, or ultraviolet light.

An ambulatory performance status of 0,1,2 (ECOG Scale).

Ability to participate in an out -patient study and to provide informed consent.

Creatinine less than 2.0 mg/100ml. Bilirubin less than or equal to 1.5 mg/100ml; prothrombin time less than or equal to 1.3 times control. WBC greater than 3000/mm(3), granulocytes greater than 1500/mm(3), platelets greater than 100,000/mm(3).

No clinically significant cardiac disease.

No patients with previously documented serious infectious diseases such as pneumocystis pneumonia, mycobacterium avium infection, etc. which would suggest clinically evident immunodeficiency.

No systemic treatment for psoriasis (methotrexate, PUVA, UVB, cyclosporine, etc.) and topical treatments (corticosteroids, tar, anthralin, etc.) during the four weeks prior to study entry, and topical treatment during the two weeks prior to study entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 1993-12; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States